CLINICAL TRIAL: NCT00798954
Title: A Multi-center Trial to Evaluate Paclitaxel- and Sirolimus-eluting Stents in Provisional T-stenting With Kissing Balloon Technique in the Treatment of Bifurcation Lesions
Brief Title: Treatment of Bifurcation Lesions by SINGLE STENT and KISSing Balloon Trial
Acronym: SINGLEKISS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Vulnerable Plaque Society (Network)
Responsible Party: Kenya Nasu, Toyohashi Heart Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SKT
Record Dates: First submitted 2008-02-12; First posted 2008-11-27 (Estimated); Last update posted 2010-06-10 (Estimated); Status verified 2010-06

CONDITIONS: Ischemic Heart Disease; Restenosis
MeSH Terms: conditions — Myocardial Ischemia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TAXUS (Active Comparator)
  Interventions: Device: Paclitaxel-eluting stent (TAXUS)
- Cypher (Active Comparator)
  Interventions: Device: Sirolimus-eluting coronary stent (Cypher)

INTERVENTIONS:
Device: Sirolimus-eluting coronary stent (Cypher) — Drug eluting stents: Comparison Sirolimus with Paclitaxel eluting stents for treatment of coronary bifurcation lesions.
  Arms: Cypher
Device: Paclitaxel-eluting stent (TAXUS) — Drug eluting stents: Comparison Sirolimus with Paclitaxel eluting stents for treatment of coronary bifurcation lesions.
  Arms: TAXUS

SUMMARY:
The use of DES have not diminished the need of improved treatment strategies , especially the treatment of bifurcation lesions still leave much to be clarified. Particularly, for bifurcation lesions where stenting the main branch could result in an obstruction of a vital side branch, many reports have been about using 2 drug-eluting stents. Resulting in less than favorable, target lesion revascularization (TLR) rates, with 10-15% for main branch and 11-40% for side branch.

In Japan, the PERFECT multi-center registry evaluated outcomes of single stenting plus kissing balloon technique after Directional Coronary Atherectomy (DCA) removal of tissue plaques. TLR rates for both main branch and side branch were a satisfactory 1.3%. However, the DCA technique is mainly suitable for proximal coronary artery lesions, and takes skilled operators.

For the treatment of relatively distal bifurcation lesions, where first POBA is performed, then the lesion is stented, followed by kissing balloon technique to fully expand the side branch, is considered a viable treatment. The Toyohashi Heart Center outcomes from August 2004 for this single stent and kissing ballooning technique, using the sirolimus-eluting stent on bifurcation lesions, achieved a satisfactory 5.2% TLR for both main and side branches, suggesting that using two stents may not be necessarily the ideal treatment.

The paclitaxel-eluting stent is expected to become available in Japan from June 2007. This stent's cells can be expanded to a maximum of 3.5mm, which should provide a larger lumen access for side-branch treatment.

As such, we developed this study to compare the outcomes of paclitaxel-eluting and sirolimus-eluting stents in bifurcation lesions that require side branch dilatation using the kissing ballooning technique.

DETAILED DESCRIPTION:
1. Primary Endpoints Target lesion revascularization after one year
2. Secondary Endpoints Secondary endpoints be evaluated in terms of safety and efficacy.

2-1 Safety

1. Major complications associated with procedure (death, QMI, CABG)
2. Major complications at follow-up (within 9 months) (death, QMI, CABG)
3. Target vessel revascularization (TVR) performed within 9 months 2-2 Efficacy

1. Acute angiographic success

* Minimum lumen diameter (MLD)

  ・% stenosis 2. Angiographic success at follow-up
* Minimum lumen diameter (MLD)

  ・% stenosis
* Loss index
* Late loss

ELIGIBILITY:
Inclusion Criteria:

Patient Inclusion Criteria:

1. Age ≥18 to <81 years and are able to undergo CABG
2. Females who are not pregnant
3. Patients who present with angina symptoms or myocardial ischemia
4. Patients available for post-procedural observation and coronary angiography at 9 months
5. Patients who have signed patient informed consent

Angiographic Inclusion Criteria:

1. Bifurcation lesion with ≥2.0mm side branch diameter as confirmed angiographically (the Duke Classification (see Reference 1)
2. The target lesion without remote lesions in the same vessel.
3. De novo lesion or non-stented restenosed lesion
4. Lesion which is eligible for stent implantation
5. Main branch reference vessel diameter of ≥2.5 mm by visual assessment
6. If two or more bifurcated lesions are present in the reference lesion, the proximal lesion shall be included in this study.

Exclusion Criteria:

Patient Exclusion Criteria:

1. Patients contraindicated for antiplatelet therapy or anticoagulant therapy
2. Patients with significant allergic reaction to contrast medium
3. Patients who are pregnant or may be pregnant
4. Patients with left ventricle ejection fraction of <30%
5. Patients deemed inappropriate by physician

Angiographic Exclusion Criteria:

1. Main branch reference vessel diameter of ≥4.5 mm by angiography
2. Bypass grafts lesions
3. In-stent restenosis lesions
4. Highly tortuous lesions of ≥60 degrees
5. Highly calcified lesions in which full stent dilatation may not be possible
6. The target lesion with remote lesions in the same vessel.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2007-06; Primary Completion 2008-12 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Target lesion revascularization | one year

CONTACTS AND LOCATIONS:
Overall Officials: Kenya Nasu, MD, Principal Investigator — Toyohashi Heart Center; Yuji Oikawa, MD, Principal Investigator — Cardiovascular Institute hospital
Locations (17):
- Japan (17):
  - Higashi Cardiovascular Clinic, Toyohashi, Aichi-ken
  - Vulnerable Plaque Society, Toyohashi, Aichi-ken
  - Toyohashi Heart Center, Toyohashi, Aichi-ken
  - Teikyo University Chiba Medical Center, Ichihara, Chiba
  - Southen Tohoku Research Institute, Kōriyama, Fukushima
  - Gunma Cardiovascular Center, Maebashi, Gunma
  - Kihara Junkanki Hospital, Asahikawa, Hokkaido
  - Chitose City Hospital, Chitose, Hokkaido
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - Shinko Kagogwa Hospital, Kakogawa, Hyōgo
  - Sanda City Hospital, Sanda, Hyōgo
  - Rinku General Medical Center, Izumisano, Osaka
  - Matsubara Tokushukai Hospital, Matsubara, Osaka
  - Tokyo Metropolitan Police Hospital, Chiyoda City, Tokyo
  - Tokyo Medical University Hospital, Shinjuku, Tokyo
  - Itabashi Chuo Medical Center, tabashi City, Tokyo
  - Cardiovascular Institute Hospital, Minatoku, Tokyou